CLINICAL TRIAL: NCT01720004
Title: Repeated Hands-and-Knees Positioning During Labour: A Pilot Randomized Controlled Trial
Brief Title: A Pilot Randomized Controlled Trial of Repeated Hands-and-Knees Positioning During Labour
Acronym: LPT2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Ellen Hodnett, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IGO-103690
Record Dates: First submitted 2012-10-24; First posted 2012-11-01 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Pregnancy, Childbirth and the Puerperium
Keywords: human labour; hands-and-knees positioning; pilot trial

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Repeated Use of Hands-and-Knees (Experimental): The intervention was repeated use of hands-and-knees position during labour. Participants were asked to try it for at least 15 minutes every hour, from randomization until delivery. They were not required to use it for delivery.
  Interventions: Other: Repeated hands-and-knees positioning during labour
- Usual care (No Intervention): Participants were asked to refrain from using hands-and-knees position at any time from randomization to delivery. They were free to use any other position.

INTERVENTIONS:
Other: Repeated hands-and-knees positioning during labour — Details are in the Arm Description.
  Arms: Repeated Use of Hands-and-Knees

SUMMARY:
The investigators designed a pilot randomized controlled trial to assess the feasibility and acceptability of repeated hands-and-knees positioning during labour. The objectives were 1) to provide an estimate of enrollment rates, 2) to assess compliance with the study protocol by participants and care providers, 3) to obtain women's views about their experiences using the hands-and-knees position, and 4) to provide estimates of treatment effects to inform the sample size calculation for a large trial.

DETAILED DESCRIPTION:
Women were enrolled in the pilot randomized controlled trial at two hospitals, one in Canada and one in the USA. Nurses at both hospitals were trained in how to assist women into the hands-and-knees position in bed. Repeated hands-and-knees position was defined as attempts to use the position for 15 minutes, hourly from randomization until delivery. Women were not asked to assume hands-and-knees for delivery.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous;
* >37 weeks 0 days gestation
* in established early labour
* anticipating a vaginal delivery of a single fetus in the cephalic position
* competent to give informed consent .

Exclusion Criteria:

* delivery was anticipated within 3 hours
* a medical contraindication or physical limitation such that hands-and- knees position was contraindicated
* had a doula or midwife who encouraged the use of hands-and-knees position.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Compliance | from randomization to delivery
  Use of hands-and-knees position for at least 15 minutes hourly during hospital labour.

SECONDARY OUTCOMES:
Persistent back pain | hourly during labour, from randomization to delivery
  Persistent back pain intensity rating measured hourly during hospital labour.
women's views | assessed prior to hospital discharge
  women's views of their birth experiences, including satisfaction with care and care providers, views about hands-and-knees positioning, willingness to use hands-and-knees position in a subsequent labour, comparison of expectations versus experiences of labour. The measures used to assess women's views had been developed for and used in prior trials of forms of intrapartum care by Hodnett and colleagues. Most questions were Likert scales or categorical items.

OTHER OUTCOMES:
Method of birth | at delivery
  Spontaneous vaginal, assisted vaginal (vacuum or forceps), Caesarean
pharmacologic analgesia | Initiated during labour
  regional analgesia or intramuscular analgesia administered during first or second stage labour
oxytocin during first or second stage labour | from randomization until end of second stage
  any oxytocin infusion
dislodged epidural catheter | from randomization until delivery
  dislodged epidural catheter
Fall | from randomization until delivery
  Mother fell while attempting hands-and-knees position
perineal trauma | at delivery
  any perineal trauma (episiotomy and/or laceration0 requiring suturing
maternal postpartum complications | between delivery and hospital discharge
  postpartum hemorrhage or complication requiring prolonged stay
Apgar Score | at one and five minutes after birth
  Neonatal Apgar Score
length of hospital stay | from delivery to discharge
  length of stay for mother and baby after birth
admission to neonatal intensive care unit | between birth and hospital discharge
  newborn admitted to neonatal intensive care unit
labour length | from randomization until delivery
  Length of time between randomization and delivery

CONTACTS AND LOCATIONS:
Locations (2):
- Texas Health Harris Methodist Hospital, Fort Worth, Texas, United States
- Toronto East General Hospital, Toronto, Ontario, Canada